CLINICAL TRIAL: NCT05277402
Title: A Phase 1b, Open-Label, Dose Escalation Study of ADG116 in Combination With Pembrolizumab (Anti-PD-1 Antibody) in Patients With Advanced/Metastatic Solid Tumors
Brief Title: ADG116 in Combination With Pembrolizumab in Patients With Advanced/Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adagene Inc (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADG116-P001; KEYNOTE-C97/MK-3475-C97 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-02-09; First posted 2022-03-14 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Advanced/Metastatic Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): ADG116 combination treatment with pembrolizumab (KEYTRUDA®), both drugs will be administered in each cohort.
  Interventions: Drug: ADG116

INTERVENTIONS:
Drug: ADG116 — IV infusion
  Other Names: Pembrolizumab (KEYTRUDA®)

SUMMARY:
This is a Phase 1b, open-label, dose escalation study to evaluate the safety, tolerability, PK, and immunogenicity of an ADG116-pembrolizumab combination regimen in patients with advanced/metastatic solid tumors. Study drug ADG116, is an anti -CTLA-4 fully human monoclonal antibody that specifically binds to human CTLA-4. Pembrolizumab is a PD-1 receptor-blocking antibody (a humanized IgG4 monoclonal antibody) which is indicated for the treatment of patients across a number of indications. The treatment strategy of using anti-PD 1 therapy combined with anti-CTLA-4 therapy is to explore the potential of combination checkpoint inhibition regimens for the enhanced antitumor efficacy results.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

  1. ≥ 18 years of age at the time of informed consent.
  2. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 with no deterioration over the previous 2 weeks.
  3. Patients with advanced or metastatic solid tumors, histologically or pathologically confirmed, who have progressed after all standard therapies, or for whom no further standard therapy exists. Patients who have declined standard therapy or have no access to standard therapy may be enrolled and the reasons for lack of access need to be documented.
  4. Patients should have at least 1 measurable lesion at baseline according to the definition of RECIST v1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
  5. Patients previously treated with anti-CTLA 4 checkpoint inhibitors or anti programmed cell death 1 (PD-1)/L1 will also be recruited if they meet all eligibility criteria. For anti-PD-1/L1 patients, patients must have progressed on treatment with an anti PD 1/L1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. Anti PD-1/L1 treatment progression is defined by meeting all of the following criteria:

     1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
     2. Has demonstrated disease progression (PD) after PD-1/L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented PD, in the absence of rapid clinical progression.
     3. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.

     i. Progressive disease is determined according to iRECIST. ii. This determination is made by the Investigator. Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression.
  6. Adequate hematologic function, defined by the following:

     1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, without the use of granulocyte colony stimulating factor such as filgrastim within 2 weeks prior to study treatment.
     2. Platelet count ≥ 100 × 109/L without transfusion within 2 weeks (≤ 14 days) prior to study treatment.
     3. Hemoglobin ≥ 9 g/dL without transfusion or erythropoietin within 2 weeks (≤ 14 days) prior to study treatment.
  7. Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN), and total bilirubin ≤ 1.5 × ULN. Exceptions: Patients who have serum bilirubin increases due to documented underlying Gilbert's Syndrome or familial benign unconjugated hyperbilirubinemia may be enrolled. Patients with known liver metastases or patients with hepatocellular carcinoma may be enrolled with AST, ALT, and/or total bilirubin ≤ 5 × the ULN.
  8. Adequate renal function defined by either a creatinine clearance ≥ 45 mL/min (by Cockcroft-Gault formula) or serum creatinine (SCr) ≤ 1.5 × ULN
  9. Coagulation tests, defined by the following:

     1. Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.
     2. International normalized ratio (INR) ≤ 1.5 × ULN. Exception: INR 2 to ≤ 3 × ULN is acceptable for patients on Warfarin anticoagulation.
  10. Left ventricular ejection fraction (LVEF) ≥ 50% measured by multiple-gated acquisition (MUGA) or echocardiogram (ECHO.).
  11. Previous antitumor therapy (including endocrine, chemoradiotherapy/ radiotherapy, targeted therapy, or immunotherapy) that has ended at least 4 weeks prior to administration of ADG116. Focal radiation therapy for symptom relief must have been completed at least 2 weeks prior to the first dose of ADG116. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease. Exception: hormonal therapy for prostate cancer is allowed (Section 6.7).
  12. Previous AEs have been improved to baseline or Grade ≤ 1 NCI CTCAE v5.0 (except for patients with alopecia). Participants with Grade ≤ 2 neuropathy may be eligible. Participants with endocrine-related AEs Grade ≤ 2 requiring treatment or hormone replacement may be eligible.

Exclusion Criteria:

* Patients who meet any of the following criteria cannot be enrolled:

  1. Pregnant or breastfeeding females.
  2. Females of childbearing potential and males whose partners are of childbearing potential who do not agree to the use of 2 forms of highly effective contraception during the treatment period and for 6 months after the last dose of study drug.
  3. Treatment with any investigational drug within 4 weeks prior to the first dose of study drug.
  4. Grade ≥ 3 immune-related AEs (irAEs) or irAE that lead to discontinuation of prior immunotherapy.
  5. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
  6. History of severe hypersensitivity (Grade ≥ 3) or known to be allergic to protein drugs or recombinant proteins or any ingredients contained in the ADG116 or pembrolizumab drug formulation.
  7. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
  8. Patients requiring systemic treatment with corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive medications within 21 days before the planned first dose of study drug. Ophthalmologic, nasal, inhaled and intra-articular injections of steroids are allowed.
  9. Patients receiving granulocyte colony stimulating factor (G-CSF), granulocyte macrophage colony stimulating factor (GM-CSF), erythropoietin, or blood (red blood cell [RBC] or platelet) transfusion within 14 days prior to the first dose of the study drug.
  10. Any evidence of underlying liver dysfunction due to other causes; Any history of significant alcohol abuse, alcoholic or drug-induced hepatitis, or documented nonalcoholic steatohepatitis.
  11. Active viral (any etiology) hepatitis patients are excluded. Hepatitis B virus (HBV) carriers are ineligible. Cured Hepatitis C (HCV) (negative HCV ribonucleic acid [RNA] test) patients may be enrolled after consulting with the Medical Monitor.
  12. Any uncontrolled active infections requiring systemic antimicrobial treatment (viral, bacterial, or other), or uncontrolled or poorly controlled diabetes as evidenced by Screening (baseline) HbA1c≥ 7.5, asthma, chronic obstructive pulmonary disease (COPD), or other conditions that pose a risk to the patient participating on study.
  13. Has a known history of HIV infection.
  14. Patients with any type of primary immunodeficiency or autoimmune disorder requiring treatment.
  15. Major surgery within 4 weeks prior to the first dose of the study drug.
  16. Has had an allogeneic tissue/solid organ transplant.
  17. Clinically significant cardiac conditions, including myocardial infarction within the last 6 months, uncontrolled angina, viral myocarditis, pericarditis, cerebrovascular accident, or other acute uncontrolled heart disease <3 months prior to the first dose of the study drug; LVEF <50%, New York Heart Association (NYHA) Class III or IV congestive heart failure, or uncontrolled hypertension.
  18. Patients with underlying hemoglobinopathies (e.g., thalassemia) will be excluded.
  19. Pulmonary embolism or deep vein thrombosis within 3 months prior to the first dose of study drug.
  20. Has received a COVID-19 vaccine within 7 days prior to the first dose of study treatment. Has received any other live or live-attenuated vaccine within 30 days prior to the first dose of study treatment. Note: Administration of killed vaccines are allowed.
  21. Has received a positive COVID-19 test within 14 days of Cycle 1 Day 1.
  22. Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
  23. Any known, documented, or suspected history of illicit substance abuse.
  24. Any other disease or clinically significant abnormality in laboratory parameters, including serious medical or psychiatric illness/condition, which in the judgment of the Investigator might compromise the safety of the patient or integrity of the study, interfere with the patient participation in the trial or compromise the trial objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) and RP2D of ADG116 in combination with pembrolizumab. | 9 months
  Number of participants experiencing dose-limiting toxicities escalating dose levels in adults with advanced / metastatic solid tumor
The safety and tolerability of ADG116 in combination with pembrolizumab | 9 month
  Number of participants with adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile/parameters | 9 Months
  Area under the time concentration curve (AUC) from time zero to infinity (AUC0-inf)
Maximum (peak) plasma concentration (Cmax) | 9 months
  Maximum (peak) plasma concentration (Cmax)
Time to maximum (peak) concentration (Tmax) | 9 month
  Time to maximum (peak) concentration (Tmax) Time to maximum (peak) concentration (Tmax)
Trough concentration (Ctrough) | 9 months
  Trough concentration (Ctrough)

CONTACTS AND LOCATIONS:
Overall Officials: Jiping Zha, MD, Study Chair — Adagene Inc
Locations (2):
- United States (2):
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Next Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No